CLINICAL TRIAL: NCT05377996
Title: A Phase 1, First-in-human, Dose Escalation and Expansion, Multicenter Study of XMT-1660 in Participants With Solid Tumors
Brief Title: A Study of XMT-1660 in Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER-XMT-1660-1
Record Dates: First submitted 2022-05-02; First posted 2022-05-17 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer; Endometrial Cancer; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XMT-1660 (Experimental): Single arm XMT-1660 alone (monotherapy)
  Interventions: Drug: XMT-1660

INTERVENTIONS:
Drug: XMT-1660 — XMT-1660 will be administered through a vein in your arm or port catheter (intravenously)

SUMMARY:
A Study of XMT-1660 in Solid Tumors

DETAILED DESCRIPTION:
This first-in-human (FIH) study will test the safety and side effects of a drug called XMT-1660. A side effect is anything a drug does to the body besides treating the disease.

Participants in the study will have cancer that has come back after a period of time during which the cancer could not be detected (recurrent), spread in the body near where it started (advanced) or spread through the body (metastatic).

The study will have two parts. The first part called Dose Escalation will find out how much XMT-1660 should be given to participants. The second part called Dose Expansion will use the dose found in the first part to find out how safe XMT-1660 is and if it works to treat solid tumor cancers.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or advanced solid tumor and has disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participants in DES must have at least one non-target lesion as defined by RECIST version 1.1. Participants in Backfill Cohorts and EXP must have at least one measurable disease (target) lesion as defined by RECIST version 1.1.
* Tumor tissue, either archival or from a fresh tumor biopsy, available for testing or be willing to undergo a minimally invasive tumor biopsy to obtain tumor tissue for local testing, if not medically contraindicated, prior to Cycle 1 Day 1
* Brain magnetic resonance imaging (MRI) during the Screening period unless obtained within 30 days prior to Screening (based on standard clinical care), if they meet either of the following criteria:

  1. All participants with TNBC
  2. Participants with a history of brain metastases or with neurologic symptoms or signs suspicious for brain metastases.

Exclusion Criteria:

* Prior treatment with an Antibody Drug Conjugate (ADC) containing an auristatin payload. Prior treatment with another ADC containing other payloads is allowed.
* Major surgery within 28 days of starting study treatment, systemic anticancer therapy within the time period of 28 days or 5 half-lives of the prior therapy before starting study treatment (14 days or 5 half-lives for small molecule targeted therapy), whichever is less, or palliative radiation therapy to the chest within 3 months of starting study treatment or to other anatomic sites within 14 days of starting study treatment.
* Diagnosis of additional malignancy that required active treatment (including surgery, systemic therapy, and radiation) within 2 years prior to screening, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix.
* Untreated CNS metastases (including new and progressive brain metastases), history of leptomeningeal metastasis or carcinomatous meningitis.
* Prior B7-H4 targeted treatment.
* History of cirrhosis, hepatic fibrosis, esophageal or gastric varices, or other clinically significant liver diseases.
* Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary, or metabolic disease) or intercurrent illness that could increase the risk of serious adverse events (SAEs) or interfere with per-protocol evaluations, in the judgment of either the Sponsor or the Investigator.
* Clinically significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events that are considered dose-limiting toxicities (DLTs) and associated with XMT-1660 during the first cycle of treatment (Dose Escalation) | 17 months
  Determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of XMT-1660
Incidence of adverse events (Dose Escalation and Dose Expansion) | 3 years
  Assess the safety and tolerability of XMT-1660 by determining the number of patients with adverse events from date of first dose to 30 days post last dose
Objective Response Rate (ORR) (Dose Expansion) | approximately 3 years
  The percentage of patients with a best overall response of complete or partial response as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Dose Escalation) | Up to approximately 3 years
  The percentage of patients with a best overall response of complete or partial response as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Duration of response (DOR) (Dose Escalation and Dose Expansion) | Up to approximately 3 years
  The time from when response criteria are first met until disease progression or death in participants who achieve a complete or partial response
Time of maximum observed plasma concentration of XMT-1660 (Tmax) (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660
Maximum observed plasma concentration of XMT-1660 (Cmax) (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660
Area under the concentration-time curve of XMT-1660 (AUC) (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660
Systemic clearance of XMT-1660 (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660 by measuring the rate at which the drug is eliminated from the body
Apparent terminal elimination half-life of XMT-1660 (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660
Volume of Distribution (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660
Trough concentration of XMT-1660 (Ctrough) (Dose Expansion) | 3 years
  Assess the pharmacokinetics of XMT-1660 by measuring the lowest concentration of drug before dosing
Assess antidrug antibodies (ADA) and neutralizing antibodies (nAB) (Dose Escalation and Dose Expansion) | 3 years
  Assess the development of antidrug antibodies (ADA) and neutralizing antibodies (nAb) to XMT-1660

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, MD, Study Director — Mersana Therapeutics
Locations (26):
- United States (26):
  - Mayo Clinic Comprehensive Cancer Center, Phoenix, Arizona
  - UC Irvine Health-Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCLA, Santa Monica, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health Hospital, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York University Langone Health, New York, New York
  - ICHAN School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center Oklahoma University Health, Oklahoma City, Oklahoma
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Oncology Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Summit Cancer Centers, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toader D, Fessler SP, Collins SD, Conlon PR, Bollu R, Catcott KC, Chin CN, Dirksen A, Du B, Duvall JR, Higgins S, Kozytska MV, Bellovoda K, Faircloth C, Lee D, Li F, Qin L, Routhier C, Shaw P, Stevenson CA, Wang J, Wongthida P, Ter-Ovanesyan E, Ditty E, Bradley SP, Xu L, Yin M, Yurkovetskiy AV, Mosher R, Damelin M, Lowinger TB. Discovery and Preclinical Characterization of XMT-1660, an Optimized B7-H4-Targeted Antibody-Drug Conjugate for the Treatment of Cancer. Mol Cancer Ther. 2023 Sep 5;22(9):999-1012. doi: 10.1158/1535-7163.MCT-22-0786. PMID 37294948